CLINICAL TRIAL: NCT01950013
Title: At-home Auditory Training Clinical Trial
Acronym: Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Larry Humes, Distinguished Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1303010805; R01DC010135 (NIH)
Record Dates: First submitted 2013-08-02; First posted 2013-09-25 (Estimated); Results first posted 2019-07-02 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Presbycusis; Aging; Hearing Loss
Keywords: Presbycusis; Aging; hearing aids; hearing training
MeSH Terms: conditions — Presbycusis; Hearing Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Passive Control (No Intervention): Hearing aid alone
- Training (Experimental): Auditory Training Program. Hearing aid plus auditory training
  Interventions: Behavioral: Auditory training program
- Active control (Sham Comparator): Sham comparator: Active control. Hearing aid plus audio-book use
  Interventions: Behavioral: Sham Comparator: Active Control

INTERVENTIONS:
Behavioral: Auditory training program — Previous experiments performed under laboratory settings using a novel word-based auditory-training regimen have demonstrated substantial improvements in open-set recognition of words and sentences in noise. The current proposed study will investigate the effectiveness of the training regimen when used in a patient's home setting with their own hearing aids.
  Arms: Training
Behavioral: Sham Comparator: Active Control — This is a sham intervention in which the patient listens to audio books following the same regimen as the patients receiving the auditory training.
  Arms: Active control

SUMMARY:
The purpose of this study is to investigate the effectiveness of an auditory training program used at home with the subject's own hearing aids.

DETAILED DESCRIPTION:
The most common communication complaint of older adults with impaired hearing is that they can hear speech, but can't understand it. This is especially true where there are competing sounds in the background. Previous experiments performed under laboratory settings using a novel word-based auditory-training regimen have demonstrated substantial improvements in open-set recognition of words and sentences in noise. The current proposed study will investigate the effectiveness of the training regimen when used in a patient's home setting with their own hearing aids. All testing for the screening, baseline speech testing, training system orientation, and the outcomes portions of this project will be conducted in the Audiology Research Laboratory (ARL) of the Speech and Hearing Center located at 200 South Jordan Avenue. The use of the training program will be done at the subject's home.

Subjects will first come to the ARL for either one session for a hearing aid follow-up and instruction in the use of the training system (Session 1) or for one session for an initial screening to determine eligibility (Screening) followed then by Session 1. Subjects will then take home a training system that includes a tablet computer that has the training program loaded onto it, a portable loudspeaker, and some accessories. There will be three groups of subjects: (1) Hearing aid alone--no training (passive control); (2) Hearing aid plus auditory training (training); and (3) Hearing aid plus audio book use (active control). Total enrollment will be 45 subjects. Those subjects in the training group and active control group will complete a 6-week training period and return to the lab for outcome measures after 6 weeks of training for the primary and secondary outcome measures. The hearing aid alone group will return for the same outcome measures as the training and active control groups, but will have no intervention between these follow-up sessions.

ELIGIBILITY:
Inclusion Criteria:

* •55-79 yrs of age

  * Native English speaker

    * Having corrected vision sufficient to read 18pt font on a computer screen
    * Wearing binaural hearing aids that were fitted within the past 3 years that are the only hearing aids the subject has ever worn

Exclusion Criteria:

* The hearing aids worn by the subject will be evaluated on the subject's ears and must be functioning as required for this study; otherwise, the subject will be excluded from participation until the hearing aids have been adjusted appropriately
* asymmetrical hearing loss
* presence of dementia, Parkinson's disease, or other neurological disorder

Ages: 55 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-07; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry E Humes, PhD, Principal Investigator — Indiana University Department of Speech and Hearing Sciences
Locations (1):
- IU Department of Speech & Hearing Sciences, Bloomington, Indiana, United States

REFERENCES:
- [Derived] Humes LE, Skinner KG, Kinney DL, Rogers SE, Main AK, Quigley TM. Clinical Effectiveness of an At-Home Auditory Training Program: A Randomized Controlled Trial. Ear Hear. 2019 Sep/Oct;40(5):1043-1060. doi: 10.1097/AUD.0000000000000688. PMID 30575602

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruiting for this study began May 1, 2013 and the final follow-up session took place on February 5, 2015. Forty-five people were recruited from a previous clinical trial on hearing aids in the lab or through newspaper advertisements and flyers.
Pre-assignment Details: No changes after enrollment except that 2 subjects withdrew prior to completion--see below.
Period: Overall Study
Arm/Group | Passive Control | Training | Active Control
Started | 15 | 15 | 15
Completed | 15 | 13 | 15
Not Completed | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Passive Control | Training | Active Control | Total
Number analyzed (Participants) | 15 | 13 | 15 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.0 (7.1) | 71.9 (6.1) | 71.3 (7.5) | 71.8 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 4 | 12
  Male | 11 | 9 | 11 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 13 | 15 | 43
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 15 | 13 | 15 | 43
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Midwestern United States-southcentral Indiana.
  participants
    United States | 15 | 13 | 15 | 43

OUTCOME MEASURES:

1. Primary Outcome: Change in Connected Speech Test (CST) Score
Description: The CST is an "objective" measure of speech-understanding in noise that will be obtained when the patient's are wearing their hearing aids. The patient hears standardized recordings of the speech in noise and then reports the sentences that were heard. These are scored as percent correct. Baseline AIDED CST score was obtained prior to the intervention period and immediately following 6-week intervention. The results reflect the CHANGE in CST from pre- to post-intervention with positive numbers indicating improved speech understanding in noise following training.
Time Frame: Baseline (prior to training) and 6-weeks later (after training)
Measure: Mean (Standard Deviation); unit: percent-correct words
Arm/Group | Passive Control | Training | Active Control
Number analyzed (Participants) | 15 | 13 | 15
percent-correct words | 3.87 (11.37) | -5.84 (22.54) | -9.60 (16.9)

2. Secondary Outcome: Change in Aided Profile of Hearing Aid Performance (PHAP) Score
Description: Change in aided performance on the Profile of Hearing Aid Performance (PHAP), a self-report measure of the frequency of listening difficulties experienced by the individual. The aided PHAP scores are proportions of time difficulties encountered in various listening situations while wearing hearing aids. Low PHAP scores indicate less frequent difficulties and reflect better aided performance. The range of possible PHAP scores are 0.0 to 1.0.There are seven subscales of the PHAP and the scores reported are based on the arithmetic means of the five subscales that deal with speech communication, PHAP global. These include the following subscale scores: EC (Ease of Communication), FT (Familiar Talkers), BN (Background Noise), Reverberation (RV) and Reduced Cues (RC). Scores reported below are the CHANGE in aided PHAP global scores, baseline minus post-training.
Time Frame: Baseline (pre-training) and 6 weeks later (post training)
Measure: Mean (Standard Deviation); unit: proportion of time had difficulties
Arm/Group | Passive Control | Training | Active Control
Number analyzed (Participants) | 15 | 13 | 15
proportion of time had difficulties | -.03 (.08) | .01 (.09) | .00 (.08)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Passive Control | Training | Active Control
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/13 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/13 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/13 | 0/15

LIMITATIONS AND CAVEATS:
The findings are limited to the efficacy and effectiveness of a relatively brief (6-week, 3x/week) at-home training regimen for older adults wearing hearing aids. More training could lead to improved benefits in everyday listening.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No